CLINICAL TRIAL: NCT00016445
Title: Phase II Study of Growth Hormone in Children With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15806; UUSOM-IRB-7797-00; GENENTECH-UUSOM-IRB-7797-00
Record Dates: First submitted 2001-05-06; First posted 2001-05-07 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; disease-related problem/condition; genetic diseases and dysmorphic syndromes; quality of life; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Growth Hormone

INTERVENTIONS:
Drug: growth hormone

SUMMARY:
OBJECTIVES: I. Determine the effect of growth hormone on height, height velocity, body weight, and lean body mass in patients with cystic fibrosis.

II. Determine the effect of growth hormone on pulmonary function in these patients.

III. Determine the impact of this drug on the quality of life in these patients.

IV. Determine if the clinical response from this drug is sustained in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive growth hormone subcutaneously (SC) daily for 1 year during the first year only.

Arm II: Patients receive growth hormone SC daily for 1 year during the second year only.

Quality of life is assessed at baseline and then every 6 months for 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of prepubertal cystic fibrosis
* No colonization by Burkholderia cepacia

--Prior/Concurrent Therapy--

* No prior or concurrent insulin requirement

--Patient Characteristics--

* Hematopoietic: No hematologic disease
* Hepatic: No liver disease
* Renal: No kidney disease
* Pulmonary: Must be able to perform pulmonary function testing
* Other: No history of diabetes Must be less than 25% of normal height and/or weight for age and sex

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2001-02; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S. Hardin, Study Chair — Southwest Medical Center at Dallas
Locations (9):
- United States (9):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County, Orange, California
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Children's Medical Center - Dayton, Dayton, Ohio
  - T.L. Carey, M.D. and Associates, Tulsa, Oklahoma
  - Southwest Medical Center at Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah